CLINICAL TRIAL: NCT04988594
Title: A 12-weeks Double Blind Trial of Effects of Yogurt With Probiotics in Adults With Type 2 Diabetes Mellitus
Brief Title: Effects of Yogurt With Probiotics in Adults With Type 2 Diabetes Mellitus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Faculty of Medical Sciences, Clinical Hospital (Other)
Responsible Party: Principal Investigator, Maria Eugenia Ruiz Diaz Narvaez, Clinical Nutritionist, Faculty of Medical Sciences, Clinical Hospital
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Health Services Research
Other Study IDs: FMSParaguay
Record Dates: First submitted 2021-06-16; First posted 2021-08-03 (Actual); Last update posted 2021-08-03 (Actual); Status verified 2021-07

CONDITIONS: Type2 Diabetes
Keywords: probiotics; glucose homeostasis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Premium probiotic yogurt (Experimental): Participants receive 300 g/d of yogurt with concentrated and freeze-dried probiotic cultures for 12 weeks. Also, the nutritional recommendations of the American Diabetes Association (ADA).
  Interventions: Dietary Supplement: Lactobacillus acidophilus 207, Bifidobacterium lactis B420/205
- Conventional yogurt (Experimental): Participants receive 300 g/d of conventional yogurt for 12 weeks. Also, the nutritional recommendations of the American Diabetes Association (ADA).
  Interventions: Dietary Supplement: Lactobacillus bulgaricus and Streptococcus thermophillus
- no fermented dairy (Experimental): Participants followed the American Diabetes Association (ADA) recommendations without including fermented dairy.
  Interventions: Dietary Supplement: No culture

INTERVENTIONS:
Dietary Supplement: Lactobacillus acidophilus 207, Bifidobacterium lactis B420/205 — Cultures containing 3.7 × 10 ^ 9 CFU/mg
  Arms: Premium probiotic yogurt
Dietary Supplement: Lactobacillus bulgaricus and Streptococcus thermophillus — Cultures containing 3.7 × 10 ^ 6 CFU/mg
  Arms: Conventional yogurt
Dietary Supplement: No culture — No probiotic cultures
  Arms: no fermented dairy

SUMMARY:
The purpose of the study is to analyze the effects of the consumption of yogurt with concentrated and lyophilized probiotic cultures on the parameters associated with glucose homeostasis, inflammation and oxidative stress in patients with Type 2 Diabetes Mellitus (T2DM).

DETAILED DESCRIPTION:
After being informed about the study and the potential risks, all patients who gave their written informed consent underwent a screening period of 1 week to determine their eligibility to participate in the study. At week 0, patients who met the eligibility requirements were randomized in a double-blind manner (participant and investigator) to the American Diabetes Association (ADA) diet + yogurt with premium probiotics (300 g/d) or ADA diet + conventional yogurt (300 g/d) or ADA diet without fermented dairy.

ELIGIBILITY:
Inclusion Criteria:

* Patients with T2DM diagnosed at least one year ago.
* That they are outpatients.
* Between 25 and 65 years old.

Exclusion Criteria:

* Smoking patients.
* Lactose intolerance.
* Pregnancy or breastfeeding.
* Presence of kidney, liver, immunodeficiency, inflammatory bowel disease or thyroid disorder.
* Use of insulin, estrogen, progesterone or diuretic injections.
* Consumption of probiotic supplements two months before the start of the study

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2021-04-30 (Actual); Study Completion 2021-04-30 (Actual)

PRIMARY OUTCOMES:
Changes from baseline in parameters associated with glucose homeostasis | Baseline and week 12
  At time 0 and after 12 weeks of intervention and follow-up, it was determined in mg/dL following the protocols established for: HDL-c (high-density lipoprotein cholesterol), LDL-c (low-density lipoprotein cholesterol), triglycerides and glucose. Likewise, glycosylated hemoglobin (HbA1c in percentage) was determined.

SECONDARY OUTCOMES:
Changes in inflammatory parameters | Baseline and week 12
  At time 0 and after 12 weeks of intervention and follow-up, the high sensitivity C-reactive protein (hs-CRP) was determined in plasma in mg/dL. Likewise, interleukin-6 (IL-6) and tumor necrosis factor alpha (TNF-a) in ng/mL.
Changes in oxidative stress parameters | Baseline and week 12
  Superoxide dismutase, glutathione peroxidase and catalase (SOD, GPx, CAT, respectively) will be measured in U/mg by spectrophotometry at time 0 and after 12 weeks of intervention and follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Pablo Perez Martinez, MD, Study Director — Instituto Maimonides de Investigacion Biomedica de Cordoba, Spain; Maria Ruiz Diaz Narvaez, DN, Principal Investigator — Faculty of Medical Science, Paraguay
Locations (1):
- Instituto Maimonides de Investigacion Biomedica de Cordoba, Córdoba, Spain